CLINICAL TRIAL: NCT05058612
Title: Midodrine for the Early Liberation From Vasopressor Support in the ICU - The LIBERATE Multi-Site Study
Brief Title: Midodrine for the Early Liberation of Vasopressor Support in the ICU (LIBERATE Multi-Site)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other); Institute of Health Economics, Canada (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00112293
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Vasoplegia
Keywords: critical care medicine; intensive care; shock; midodrine
MeSH Terms: conditions — Vasoplegia; Shock | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine (Experimental): Midodrine 10 mg PO/NG q8h
  Interventions: Drug: Midodrine
- Placebo (Placebo Comparator): Microcrystalline cellulose PO/NG q8h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine — 10 mg PO/NG q8h
  Arms: Midodrine
Drug: Placebo — Microcrystalline cellulose PO/NG 18h
  Arms: Placebo

SUMMARY:
Vasopressors are medications that are given intravenously to increase the blood pressure of patients with illnesses that cause dangerous blood pressure drops. When a doctor prescribes a vasopressor, they ask that the dose be adjusted to achieve a specific blood pressure. This kind of medical support with intravenous (IV) vasopressors are usual treatments in intensive care unit (ICU) settings. Oral vasopressors, such as midodrine, have been historically used to maintain blood pressure in non-critically ill patients. In this study, the investigators will be using midodrine to reduce the need for IV vasopressors as blood pressure improves during the stay in the ICU.

This LIBERATE multi-site study will continue the work of the LIBERATE feasibility RCT study to evaluate the role of midodrine for patients with low blood pressure in the ICU. It is comprised of the multi centre pilot RCT followed by the definitive multi centre RCT.

DETAILED DESCRIPTION:
Purpose: Resuscitation and hemodynamic support with intravenous (IV) vasopressors is a prime indication of treatment in intensive care unit (ICU) settings. Hemodynamic support is typically provided with intravenous (IV) vasopressors. However, these have been shown to have significant negative effects including increased central venous catheter line associated infections, venous thromboembolic disease, impaired mobility and gastrointestinal injury and ischemia. Oral vasopressors, such as midodrine, have been historically used for hemodynamic support in non-critically ill patients, but their study in patients as IV pressor sparing therapy has been limited.

Hypothesis: to evaluate the expanded role of midodrine for any vasoplegic patients in the ICU.

Justification: In 2018, there were 1,613 admissions to the adult general systems ICU (GSICU) at the University of Alberta Hospital (UAH). Patients were sick, with a mean Acute Physiology and Chronic Health Evaluation II (APACHE) score of 21.3, with 36.4% requiring vasopressors on admission, accounting for 1942 patient-days (data from eCritical TRACER database). In the environment strained healthcare resources and limited ICU capacity, the ability to safely wean patients from IV vasopressors with transition to oral hemodynamic supporting agents would greatly improve how patients navigate through the healthcare system. This in turn will improve patient-centered case.

Primary Objective:

To compare the effect of enteral midodrine vs. placebo in critically ill patients with vasoplegia receiving continuous IV vasopressor therapy on a hierarchical composite of 28-day mortality and ICU length of stay.

Secondary Objectives: To compare the effect of enteral midodrine vs. placebo on: 28-day, hospital, and 90-day mortality, Duration of IV vasopressor support, Rates of ICU re-admission, Rate of re-initiation of IV vasopressors, and Quality of life at one year.

Tertiary Objectives: To determine the health economic effects of the usage of midodrine vs placebo on: ICU costs, Hospital costs, Total healthcare costs, Cost-effectiveness.

Safety Endpoints: Adverse drug reactions, Serious adverse drug reactions, Suspected unexpected serious adverse reactions.

Research Method/Procedures: The LIBERATE Trial is a multi center, concealed-allocation parallel-group blinded randomized controlled trial. Patients will be randomly assigned to midodrine (enteral, 10mg every 8h) or placebo (microcrystalline cellulose) for the duration of their IV vasopressor therapy and 24h following the discontinuation of their IV vasopressor therapy. The recruitment target for the multi centre pilot RCT is 350 subjects (i.e., 175 subjects per arm), followed by the definitive RCT with a recruitment target of 870 subjects (435 subjects per arm). A blinded multi site pilot analysis will be conducted after the enrolment of the first 20% of study subjects (170 subjects).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Ongoing vasopressor support
* Decreasing vasopressor dose(s)

Exclusion Criteria:

* Greater than 24 hours from peak vasopressor dose
* Contraindication to enteral medications
* Previously received midodrine in last 7 days
* Expected death or anticipated withdrawal of life-sustaining therapies in next 24 hours
* Pregnancy
* Known allergy to midodrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of 28-day mortality and ICU length of stay | 1 year
  The effects of midodrine on patient mortality at 28 days or total duration of patient stay in ICU

SECONDARY OUTCOMES:
Mortality | 1 year
  28-day, hospital and 90-day mortality
Total and post-ICU length of stay | 1 year
  The total duration of patient stay in hospital and the duration of hospital stay after ICU discharge
Duration of vasopressor support | 1 year
  Duration of intravenous vasopressor support
ICU readmission | 1 year
  Rate of ICU re-admissions during the index hospitalization
Re-initiation of vasopressors | 1 year
  Rate of re-initiation of intravenous vasopressors during ICU stay
Quality of life as measured by the EQ-5D-5L | 1 year
  The quality of life score
ICU costs | 1 year
  Total cost of ICU stay
Hospital costs | 1 year
  Total cost of hospital stay
Total health care costs | 1 year
  Total healthcare costs
Cost effectiveness | 1 year
  Incremental costs and effectiveness based on daily ICU costs

CONTACTS AND LOCATIONS:
Overall Officials: Oleksa Rewa, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Opgenorth D, Baig N, Fiest K, Karvellas C, Kutsogiannis J, Lau V, Macintyre E, Senaratne J, Slemko J, Sligl W, Wang X, Bagshaw SM, Rewa OG. LIBERATE: a study protocol for midodrine for the early liberation from vasopressor support in the intensive care unit (LIBERATE): protocol for a randomized controlled trial. Trials. 2022 Mar 4;23(1):194. doi: 10.1186/s13063-022-06115-0. PMID 35246227